CLINICAL TRIAL: NCT00240461
Title: Efficacy and Safety of COLD-fX in the Prevention of Respiratory Infections in Community-dwelling Seniors: a Multi-center, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Use of COLD-fX to Prevent Respiratory Infections in Community Dwelling Seniors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Capital Health, Canada (Other)
Collaborators: Afexa Life Sciences Inc (Industry); IWK Health Centre (Other); Sunnybrook Health Sciences Centre (Other); Erasmus Medical Center (Other); University of BC Gerontology & Diabetes Research (Other)
Responsible Party: Dr. Gerry Predy, Capital Health
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CVT-E002-2005-2
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Respiratory Tract Infection
Keywords: respiratory; infection; influenza
MeSH Terms: conditions — Respiratory Tract Infections; Infections; Influenza, Human | interventions — Dietary Supplements; COLD-fX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 200 mg COLD-fX Natural health products 2 times daily for six months
  Interventions: Dietary Supplement: COLD-fX natural health product
- Arm 2 (Active Comparator): Arm 2 - 400 mg COLD FX Natural health product - 2 times daily for 6 months
  Interventions: Dietary Supplement: COLD-fX
- 3 (Placebo Comparator): Inactive crystalline substance. This is the placebo arm in which subject receive 200 mg of the placebo 2 times daily for 6 months. Placebo is an inactive crystalline substance.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: COLD-fX natural health product — 200 mg/COLD-fX natural health product - 2 capsules twice daily for 6 months
  Other Names: Natural health product; dietary supplement
  Arms: 1
Dietary Supplement: COLD-fX — 400 mg COLD-fX natural health product 2 times daily for 6 months
  Other Names: naural health products; dietary supplements
  Arms: Arm 2
Other: Placebo — crystalline substance 200 mg twice daily for 6 months
  Other Names: none available
  Arms: 3

SUMMARY:
Seniors are a population vulnerable to respiratory infections. It is hypothesized that regular use of COLD-fX following an influenza vaccination would potentially augment immune response in the elderly. Use of COLD-fX may also provide additional protection again respiratory infection and reduce the incidence and severity of respiratory infections in otherwise healthy seniors.

DETAILED DESCRIPTION:
Eligible seniors will be randomly placed into three groups to receive 400 mg/day, 800mg/day or a placebo for a period of six months beginning in October. Daily dosing will be recorded as well as any symptoms not related to having a respiratory infection. For seniors who experience a respiratory infection, they are asked to call a study nurse who will take a nasopharyngeal swab. The seniors are also asked to record on a diary card the severity of their symptoms on a scale from 0-3 (none, mild, moderate, severe). Symptoms include cough, fever, runny nose, stuff nose, aches and pains, headache, chills, sneezing, ear aches and fatigue.The swab will be taken to the lab for testing for upper respiratory viruses.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years of age and older
* current season influenza immunization
* available for follow-up visits
* willing and able to sign written informed consent

Exclusion Criteria:

* HIV infection
* malignancy (under active observation or treatment)
* unstable cardiovascular diseases
* renal abnormalities (serum creatine >200umol/l)
* pulmonary disease (chronic bronchitis, emphysema, or asthma requiring treatment in the last 3 months with oral steroids - prednisone >10mg/day, other chronic respiratory illness)
* acute or active chronic liver disease
* neurologic or psychiatric disease (progressive or currently under treatment
* active tuberculosis
* multiple sclerosis
* bleeding disorders
* planned surgery over the course of the trial
* on immunosuppressive therapy
* taking oral steroids at dose = to prednisone 10 mg/day or more
* taking phenelzine, pentobarbital, haloperidol, warfarin, heparin
* use of natural health products(except the study product and vitamins and minerals with a dose <600 mg/day of vitamin E and containing no vitamin K) including echinacea or ginseng-containing products (tea, capsules, extracts, tablets)
* current alcohol/drug abuse
* major surgery in the past 6 months
* allergies to ginseng

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 780 (Actual)
Dates: Start 2005-09; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To determine the effects of COLD-fX supplementation on the incidence of laboratory and clinically confirmed upper respiratory infections. | During the study time frame of 6 months

SECONDARY OUTCOMES:
To evaluate the effects of the treatment on the incidence and frequency of all respiratory infections meeting the Jackson criteria and to determine the efficacy of COLD-fX supplementation on the severity and duration of symptoms. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Gerry Predy, MD, Principal Investigator — Capital Health, Canada; Shelly McNeil MD, Principal Investigator — IWK Health Centre; Jan McElhaney, Principal Investigator — UBC Gerontology and Diabetes Research; Andrew Simor MD, Principal Investigator — Sunnybrook Health Sciences Centre; Albert Osterhaus Dr., Principal Investigator — Erasmus Medical Centre
Locations (5):
- Canada (4):
  - Alberta Health Services, Edmonton, Alberta
  - UBC Gerontology and Diabetes Research, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- Dr. Albert Osterhaus, Rotterdam, Netherlands